CLINICAL TRIAL: NCT06161545
Title: A Phase II Sequential Window of Opportunity Trial of Pembrolizumab + N-803 Alone or in Combination With PD-L1 t-haNK Cells for Resectable Head and Neck Squamous Cell Carcinoma
Brief Title: Pembrolizumab + N-803 Alone or in Combination With PD-L1 t-haNK Cells for Resectable Head and Neck Squamous Cell Carcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 10001564; 001564-C
Record Dates: First submitted 2023-12-04; First posted 2023-12-08 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10-02

CONDITIONS: Stage II Squamous Cell Carcinoma of the Head and Neck; Stage III Squamous Cell Carcinoma of the Head and Neck; Stage IV Squamous Cell Carcinoma of the Head and Neck
Keywords: Anti PD-1; ALT-803; triplet; p-16 negative; HPV negative
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — pembrolizumab; ALT-803

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Experimental): N-803 + pembrolizumab
  Interventions: Drug: pembrolizumab; Drug: N-803
- Arm 2 (Experimental): N-803 + pembrolizumab + PD-L1 t-haNK cells
  Interventions: Biological: PD-L1 t-haNK cells; Drug: pembrolizumab; Drug: N-803

INTERVENTIONS:
Biological: PD-L1 t-haNK cells — Irradiated PD-L1 t-haNK cells at a dose of 2 x 10^9 administered via IV infusion over 30 minutes on Days 1, 5, 8, 12, and 15
  Arms: Arm 2
Drug: pembrolizumab — 400 mg administered as a 30 minute IV infusion on Day 1
Drug: N-803 — 15 ug/kg via subcutaneous injection on Day 1

SUMMARY:
Background:

Squamous cell carcinoma is a type of cancer that can cause tumors on the head and neck (HNSCC). Even with treatment, less than 50% of people with certain types of HNSCC survive for 5 years.

Objective:

To test a new drug treatment (N-803 and pembrolizumab, with or without PD-L1 t-haNK cells) in people with HNSCC. These drugs may help the immune system to fight cancer.

Eligibility:

People aged 18 years and older who have HNSCC that is not linked to human papillomavirus infection. They must not yet have received any treatment and be scheduled for surgery to remove the tumors.

Design:

Participants will be screened. They will have a physical exam with blood and urine tests. They will have imaging scans and a test of their heart function. They will have a biopsy: A sample of tissue will be removed from the tumor.

Pembrolizumab is given through a tube attached to a needle inserted into a vein in the arm (intravenous infusion). N-803 is injected under the skin of the abdomen. All participants will receive these 2 treatments on day 1. They will have follow-up visits on days 8 and 15.

Some participants will also receive PD-L1 t-haNK cells by intravenous infusion. These are cells that attack cancer cells. These participants will receive this treatment on days 1, 5, 8, 12, and 15.

All participants will have a clinic visit on day 21. They will have a second biopsy.

Follow-up visits will occur on days 49 and 105. Visits will continue by phone or email every 9 weeks for 2 years....

DETAILED DESCRIPTION:
Background:

* Even in the potentially curative setting, human papillomavirus (HPV)-unrelated head and neck squamous cell carcinomas (HNSCC) are associated with dismal outcomes (compared to HPV-related) despite maximal surgical and adjuvant treatment (i.e., radiotherapy +/-chemotherapy).
* The window period between diagnosis and curative surgery provides a window of opportunity to administer therapies that may improve outcomes.
* Four published clinical trials suggest that neoadjuvant checkpoint blockade can improve recurrence-free survival (RFS) in resectable HNSCC (NCT02919683, NCT02488759, NCT02296684, NCT04247282). This includes NCI protocol 20C0024 (NCT04247282) where in addition to demonstrating improved 1-year RFS compared to historical values, our correlative studies provided insight into potential mechanisms of this benefit.
* N-803 (an IL-15 agonist) combined with anti-programmed cell death protein 1 (PD-1) therapies work toward maximization of T cell-mediated anti-tumor activity, a key component of anti-tumor immunity. However, expression of T cell inhibitory receptors and/or loss of antigen presentation and processing machinery, often driven by T cell activity s release of interferon-gamma renders some tumor cells invulnerable to T cell killing.
* Studies conducted by collaborators at the NCI have shown that programmed death-ligand (PD-L1) t-haNK can lyse such T-cell-resistant tumor cells. Additionally, in a murine model of oral cancer, the triplet of PD-L1 t-haNK combined with pembrolizumab and N-803 resulted in more tumor control than the doublet combinations of these agents.
* PD-L1 t-haNK cells is an allogenic, irradiated (no engraftment), off-the-shelf cell line currently being studied in combination with pembrolizumab and N-803 in advanced/metastatic HNSCC (NCI CCR protocol 000096, (NCT04847466)). As of November 2022, 10 participants have been treated and the regimen has been well tolerated.
* In addition to potentially improving outcomes, testing this triplet in the neoadjuvant setting with pre-and post-treatment tumor biopsies provides an opportunity to gain insight into the mechanisms of this regimen s anti-tumor activity.

Objective:

-To determine the pathologic tumor response (pTR) rate (viable tumor in 50% or less of the surgically resected primary tumor bed) in Arm 1 and Arm 2

Eligibility:

* Histologically or cytologically confirmed previously untreated intermediate/high risk, p16-negative (if oropharyngeal primary tumor), squamous cell carcinoma of the head and neck (T1-T4, N0-N3, M0 stage II, III or IV.
* Age >= 18 years.
* Eastern Cooperative Oncology Group (ECOG) performance status <= 1 and adequate organ function.

Design:

* This is an open-label, single-site, non-randomized, phase II study to evaluate the efficacy of combined treatment of PD-L1 t-haNK cells, pembrolizumab, and N-803.
* The first 15 participants will be enrolled in Arm 1 and treated with pembrolizumab and N-803, the following participants will be enrolled in Arm 2 and treated with pembrolizumab, N-803, and PD-L1 t-haNK cells.
* All participants (Arm 1 and Arm 2) will receive treatment consisting of one intravenous (IV) infusion of pembrolizumab and one subcutaneous (SC) injection of N-803 on Day 1.
* Participants in Arm 2 will receive additional treatment with IV infusion of PD-L1 t-haNK cells on Days 1, 5, 8, 12, and 15.
* Participants will be monitored for 2 years.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Histologically or cytologically confirmed previously untreated intermediate/high risk, p16-negative (if oropharyngeal primary tumor), squamous cell carcinoma of the head and neck (T1-T4, N0-N3, M0 stage II, III or IV). Note: p16 status will be determined by a history of p16 immunohistochemistry (IHC) staining conducted per standard of care.
* Age >= 18 years.
* ECOG performance status <= 1.
* Planned for cancer removal surgery per standard of care.
* Participants must have adequate organ and marrow function as defined below:

  * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) <= 3.0 x upper limit of normal (ULN)
  * Total bilirubin <= 1 x ULN. Note: Participants with Gilbert's syndrome can have total bilirubin < 3.0 mg/dL
  * Absolute neutrophil count (ANC) >= 1.0 x 10^9/L
  * Hemoglobin (Hgb) >= 10.0 g/dL
  * Platelet count >= 100 x 10^9/L
  * Prothrombin time (PT) and partial thromboplastin time (PTT) <= 1 x ULN. Note: Participants with prolonged PTT determined to be due to lupus anticoagulant are eligible
  * Creatinine <= 1.5 x ULN
* Participants with a history of human immunodeficiency virus (HIV) infection must:

  * be on effective anti-retroviral therapy; and
  * have the viral load < 400 copies/mL; and
  * have the CD4 count > 150 cells/microL
* Participants with a history of Hepatitis C virus (HCV) infection must

  * received curative treatment; and
  * have an undetectable viral load.
* Individuals of child-bearing potential (IOCBP) and those who can father children must agree to use an effective method of contraception (barrier, hormonal, intrauterine device (IUD), surgical sterilization) for the duration of the study treatment and up to 4 months after the last dose of the study drug (s).
* Nursing participants must be willing to discontinue nursing from study treatment initiation through 4 months after the last dose of the study drug(s).
* Participants must have a primary tumor site that is amenable to biopsy and be willing to undergo pre-and post-treatment biopsies.
* The ability of a participant to understand and the willingness to sign a written informed consent document.

EXCLUSION CRITERIA:

* History of allergic reactions attributed to compounds of similar chemical or biological composition to drugs used in the study.
* Active immunosuppressive treatment equivalent of > 10mg of prednisone daily. Note: Short-course systemic corticosteroids (e.g., prevention/treatment for transfusion reaction) or use for a non-cancer indication (e.g., adrenal replacement) is acceptable.
* History of autoimmune disease with the exception of controlled thyroid disease, psoriasis not requiring medications, vitiligo, and alopecia.
* Participants with a history of hepatitis B (HBV).
* Prior malignancy active within the previous 2 years except for locally curable cancer that is currently considered cured and does not require an additional standard of care treatment, such as cutaneous basal or squamous cell carcinoma, superficial bladder cancer, or cervical carcinoma in situ, or an incidental histological finding of prostate cancer.
* Prior therapy with the investigational drug within 2 weeks prior to the treatment initiation.
* Pregnancy (confirmed with Beta-human chorionic gonadotropin (Beta-HCG) serum or urine pregnancy test performed in individuals of childbearing potential at screening).
* Uncontrolled intercurrent illness or medical condition(s) evaluated by medical history and physical exam or situations that are not stable (e.g., recent hospitalization, Emergency Room visit or undergoing medication changes) that the investigator assesses would unacceptably increase of participation in the trial for the participant or impair the ability to evaluate the endpoints of the study.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-09-24 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
pTR rate (viable tumor in 50% or less of the surgically resected primary tumor bed) | From enrollment to 5 days after the last infusion of PD-L1 t-hank cells or at least 20 days after pembrolizumab/N-803 administration.
  Digital pathology software assessment of H and E slides from the surgical specimen. The fraction of participants on each arm who experience a pathologic tumor response (pTR) will be reported along with a 95% confidence interval.

SECONDARY OUTCOMES:
Safety | 90 days after surgery
  Safety will be evaluated by determining the frequency of adverse events among treated participants and reporting the results, by maximum grade of event and type of toxicity noted.
Recurrence free survival | 2 years
  Determined on each arm separately using a Kaplan-Meier curve. The one-year and two-year OS and RFS will be determined and reported on each arm along with a 95% confidence interval.
Overall survival | 2 years
  Determined on each arm separately using a Kaplan-Meier curve. The one-year and two-year OS and RFS will be determined and reported on each arm along with a 95% confidence interval.
Median time from diagnosis to definitive surgery | time of surgery
  Record the date of diagnosis and date of definitive surgery. The median for each Arm will be determined.

CONTACTS AND LOCATIONS:
Overall Officials: Charalampos Floudas, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD will be shared. All IPD recorded in the medical record will be shared with intramural investigators upon request. In addition, all large scale genomic sequencing data will be shared with subscribers to dbGaP.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: This study will comply with the NIH Data Management and Sharing (DMS) Policy. Genomic data are available once genomic data are uploaded per protocol GDS plan for as long as database is active.
Access Criteria: Data from this study may be requested by contacting the PI. Genomic data are made available via dbGaP through requests to the data custodians.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_001564-C.html